CLINICAL TRIAL: NCT01290796
Title: Clinical Evaluation of Ajust™ in Stress Urinary Incontinence (CEASe)
Brief Title: Clinical Evaluation of Ajust™ in Stress Urinary Incontinence
Acronym: CEASe
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: C. R. Bard (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BMD-2112
Record Dates: First submitted 2011-02-04; First posted 2011-02-07 (Estimated); Results first posted 2014-05-12 (Estimated); Last update posted 2017-03-27 (Actual); Status verified 2017-02

CONDITIONS: Female Stress Urinary Incontinence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ajust Adjustable Single-Incision Sling (Other): Urinary incontinence sling
  Interventions: Device: Ajust Adjustable Single-Incision Sling

INTERVENTIONS:
Device: Ajust Adjustable Single-Incision Sling — The Ajust™ Adjustable Single-Incision Sling is a minimally invasive suburethral sling indicated for the treatment of female SUI resulting from urethral hypermobility and/or intrinsic sphincter deficiency (ISD). The system consists of a unique adjustable polypropylene mesh sling with permanent, self-fixating, polypropylene anchors, an introducer, and a flexible stylet for securing the mesh sling after adjustment.

SUMMARY:
The purpose of this study is to assess the overall effectiveness of the Ajust Adjustable Single-Incision Sling in the surgical treatment of female stress urinary incontinence.

DETAILED DESCRIPTION:
Urinary incontinence (UI), or the complaint of any involuntary loss of urine, ranges in severity from the occasional leaking urine during actions resulting in increased abdominal pressure (coughing, sneezing, laughing, exercise, etc.) to sudden, unpredictable strong urges to void. Female stress urinary incontinence (SUI) is attributed to a weakening of the pelvic floor muscles.

A recent review of literature describing the prevalence of UI calculated the median prevalence of female UI to be 27.6% (4.8-58.4%), with the prevalence of significant incontinence increasing with age. The prevalent cause of UI was further categorized into stress (50%), mixed (32%) and urge (14%).

Nonsurgical treatment of female SUI has traditionally been limited to alpha-adrenergic agonists and estrogens, pelvic floor exercises, biofeedback, electrical stimulation and behavior modification1. Options for surgical treatment consists of periurethral injections of bulking agents, transvaginal suspensions, retropubic suspensions, slings and sphincter prostheses.

The Ajust™ Adjustable Single-Incision Sling is a fully adjustable single-incision sling that anchors in the transobturator membranes, anatomically sufficient spaces for support of the urethra.

ELIGIBILITY:
Inclusion Criteria:

* Female, age at least 18 years
* Have signed an Informed Consent Form
* Has been diagnosed with stress urinary incontinence as documented by: a minimum 30-degree urethral deflection, considered to be a candidate for transobturator repair by consulting surgeon (investigator), has a positive CST
* Desires surgical correction of SUI using the Ajust™ Adjustable Single-Incision Sling

Exclusion Criteria:

* Patient is actively participating in any other genitourinary clinical trial of an experimental drug or device
* Patient is known to be pregnant or desiring future childbearing
* Patient has a known urinary tract infection, or known infection in the operative field at the time of device implantation
* Patient is unable to have their anticoagulation therapy suspended for the completion of the surgical procedure
* Patient requires concurrent correction of pelvic organ prolapse
* Patient has a history of previous sling procedure
* Patient has known history of detrusor overactivity demonstrated by urodynamics
* Patient has known urinary retention
* Patient has a current genitourinary fistula or urinary diverticulum
* Patient has a prior history of pelvic radiation
* Patient has a MESA urge symptom score (% of total possible urge score) that is greater than their MESA stress symptom score (% of total possible stress score)
* Any condition in the opinion of the Investigator that would preclude the use of the Ajust™ Adjustable Single-Incision Sling, or preclude the subject from completing the follow-up requirements

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 153 (Actual)
Dates: Start 2011-01; Primary Completion 2013-06 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Lucente, MD, Principal Investigator — Institute for Female Pelvic Medicine and Reconstructive Surgery
Locations (6):
- United States (6):
  - Clark Center for Urogynecology, Newport Beach, California
  - Female Pelvic & Urogynecology Institute of Michigan, Grand Rapids Womens Health, Grand Rapids, Michigan
  - Princeton Urogynecology, Princeton, New Jersey
  - Institute for Female Pelvic Medicine and Reconstructive Surgery, Allentown, Pennsylvania
  - Manjon Gynecology, Harrisburg, Pennsylvania
  - Southern Uroynecology, West Columbia, South Carolina

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ajust Adjustable Single-Incision Sling
Started | 153
Completed | 123
Not Completed | 30
Not completed — Lost to Follow-up | 21
Not completed — Withdrawal by Subject | 4
Not completed — Physician Decision | 2
Not completed — Secondary Surgical Intervention | 2
Not completed — Withdrawal by Sponsor | 1

BASELINE CHARACTERISTICS:
Arm/Group | Ajust Adjustable Single-Incision Sling
Number analyzed (Participants) | 153
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.4 (10.3)
Age, Customized [Number; unit: participants]
  <65 years | 129
  >=65 years | 24
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 153
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 5
  Native Hawaiian or Other Pacific Islander | 2
  Black or African American | 3
  White | 143
  More than one race | 0
  Unknown or Not Reported | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 149
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 153

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients Free of Stress Urinary Incontinence
Description: Percentage of patients who are free of stress urinary incontinence, as assessed by a negative (-) Cough Stress Test (CST) and no surgical retreatment, at the 12 month study visit.
Time Frame: 12-months post surgical procedure
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ajust Adjustable Single-Incision Sling
Number analyzed (Participants) | 153
percentage of participants | 92.8 [87.1 to 96.5]

2. Primary Outcome: Percentage of Subjects Who Showed Improvement in Self-reported SUI Symptoms at 12 Months
Description: Improvement was defined as a 25-point decrease (improvement) in Urinary Distress Inventory (UDI-6) score (Range: 0 - 100).
Time Frame: 12-months post procedure
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ajust Adjustable Single-Incision Sling
Number analyzed (Participants) | 153
percentage of participants | 79.3 [71.4 to 85.8]

3. Secondary Outcome: Operative, Perioperative and Long-Term Complications During Operative Procedure
Description: Percentage of Patients with Procedure and/or Device Related Adverse Events During the Operative Procedure
Time Frame: 1 day
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ajust Adjustable Single-Incision Sling
Number analyzed (Participants) | 153
percentage of participants | 11.8 [7.1 to 18.0]

4. Secondary Outcome: Operative, Perioperative and Long-Term Complications Perioperatively
Description: Percentage of Patients with Procedure and/or Device Related Adverse Events Perioperatively
Time Frame: 1-15 days
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ajust Adjustable Single-Incision Sling
Number analyzed (Participants) | 153
percentage of participants | 2.6 [0.7 to 6.6]

5. Secondary Outcome: Operative, Perioperative and Long-term Complications Through 36 Months
Description: Percentage of Patients with Procedure and/or Device Related Adverse Events through 36 months
Time Frame: Day 15 through 36-months post procedure
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ajust Adjustable Single-Incision Sling
Number analyzed (Participants) | 153
percentage of participants | 8.5 [4.6 to 14.1]

6. Secondary Outcome: Change in Post-operative Pain
Description: Mean change in Overall McCarthy Surgical Pain Scale from Day 0 to Day 7. McCarthy Pain Scale is a 50 millimeter line with "No Pain Sensation" noted at the 0 mm mark and "Most Intense Pain Imaginable" noted at the 50 mm mark. Each day, subjects are asked to mark their level of pain somewhere along the line. Change in pain level is reported in millimeters.
Time Frame: 0-7 days
Measure: Mean (Standard Deviation); unit: millimeters
Arm/Group | Ajust Adjustable Single-Incision Sling
Number analyzed (Participants) | 153
millimeters | -79.7 (92.7)

7. Secondary Outcome: Percentage of Subjects Who Showed Improvement in Self-reported SUI Symptoms at 36 Months
Description: as for outcome 2
Time Frame: 0-36 Months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ajust Adjustable Single-Incision Sling
Number analyzed (Participants) | 153
percentage of participants | 55.3 [46.1 to 64.3]

8. Secondary Outcome: Change in Incontinent Impact Questionnaire at 12 Months
Description: Mean change in overall IIQ-7 summary score (range 0 - 100). Scores on the IIQ-7 range from 0 (best outcome) to 100 (worst outcome). For this outcome measure, IIQ-7 at baseline was compared to that administered at 12-months post-surgery.
Time Frame: 0-12 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ajust Adjustable Single-Incision Sling
Number analyzed (Participants) | 153
units on a scale | -32.9 (23.5)

9. Secondary Outcome: Change in Incontinent Impact Questionnaire at 36 Months
Description: Mean change in overall IIQ-7 summary score (range 0 - 100). Scores on the IIQ-7 range from 0 (best outcome) to 100 (worst outcome). For this outcome measure, IIQ-7 at baseline was compared to that administered at 36-months post-surgery.
Time Frame: 0-36 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ajust Adjustable Single-Incision Sling
Number analyzed (Participants) | 153
units on a scale | -29.7 (22.2)

10. Secondary Outcome: Percentage of Patients With Impression of Improvement With Procedure at 12 Months
Description: Patient satisfaction was assessed using the Patient Global Impression of Improvement (PGII) questionnaire. Patients were considered to be "satisfied" if they felt that their urinary tract condition was "very much better" or "much better" than how it felt before the surgery.
Time Frame: 0-12 Months
Population: Patients who completed 12 month evaulations
Measure: Number; unit: percentage of participants
Arm/Group | Ajust Adjustable Single-Incision Sling
Number analyzed (Participants) | 136
percentage of participants | 94.9

11. Secondary Outcome: Percentage of Patients With Impression of Improvement With Procedure at 36 Months
Description: Patient satisfaction was assessed using the Patient Global Impression of Improvement (PGII) questionnaire. Patients were considered to be "satisfied" if they felt that their urinary tract conditio0n was "very much better" or "much better" than how it felt before the surgery.
Time Frame: 0-36 Months
Population: Patients who completed 36 month evaulations
Measure: Number; unit: percentage of participants
Arm/Group | Ajust Adjustable Single-Incision Sling
Number analyzed (Participants) | 123
percentage of participants | 81.3

ADVERSE EVENTS:
Arm/Group | Ajust Adjustable Single-Incision Sling
Serious Adverse Events (participants affected / at risk) | 2/153
Other Adverse Events (participants affected / at risk) | 16/153
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ajust Adjustable Single-Incision Sling (N=153)
Anuria (Renal and urinary disorders) | 1 (1)
Implant Site Pain (General disorders) | 1 (1)
Medical device complication (Injury, poisoning and procedural complications) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ajust Adjustable Single-Incision Sling (N=153)
Procedural Pain (Injury, poisoning and procedural complications) | 16 (16)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No